CLINICAL TRIAL: NCT06909266
Title: Impact of Vestibular Function on Deaf Infants' Activities of Daily Living
Acronym: IVANS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250135; IDRCB: 2025-A00243-46 (Registry Identifier: ANSM)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Dysfunction; Hearing Loss; Motor Development
Keywords: Deafness; vestibular disorder; occupational therapy
MeSH Terms: conditions — Hearing Loss; Deafness; Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- deaf children with vestibular disorder: Children aged 0 to 2 years old
  Interventions: Other: OT Hope 0 - 5 ans Therapeutic tool; Other: Qualitative interviews with parents
- deaf children without vestibular disorder: Children aged 0 to 2 years old
  Interventions: Other: OT Hope 0 - 5 ans Therapeutic tool; Other: Qualitative interviews with parents
- hearing children without vestibular disorder: Children aged 0 to 2 years old
  Interventions: Other: OT Hope 0 - 5 ans Therapeutic tool; Other: Qualitative interviews with parents

INTERVENTIONS:
Other: OT Hope 0 - 5 ans Therapeutic tool — OT Hope 0 - 5 ans Therapeutic tool for self determination of pediatric goals in occupational therapy
Other: Qualitative interviews with parents — qualitative interviews to understand how vestibular impairments affect their child's daily life activities, challenges encountered, and strategies used to support participation.

SUMMARY:
This non-interventional study aims to assess the impact of vestibular impairments on the daily life activities of deaf children aged 0 to 2 years old. Three groups of participants will be included: deaf children with vestibular impairment, deaf children without vestibular impairment, and hearing children without vestibular dysfunction (control group).

Children's daily activities will be evaluated through the OT Hope 0-5 years tool, a parent-administered questionnaire designed to measure competencies in different areas: personal care, play, and social interactions. This study also includes qualitative interviews with parents to further explore how vestibular impairments affect children's daily routines.

It is hypothesized that:

* Deaf children with vestibular impairments will show lower scores in daily life activities compared to the other two groups.
* Deaf children without vestibular impairments will demonstrate scores closer to those of hearing children but may show some differences due to their hearing status.

The research is conducted at the Robert Debré Hospital, in Paris, and aims to enroll 105 children over a three-year period. The data collected will provide insights into the specific needs of children with vestibular impairments and lay the groundwork for targeted early interventions.

DETAILED DESCRIPTION:
This non-interventional, observational, case-control study aims to evaluate the impact of vestibular impairments on the daily life activities and functional development of deaf children aged 0 to 2 years. The study focuses on understanding how vestibular dysfunction, a condition affecting balance, posture, and motor skills, influences children's ability to perform essential daily tasks such as walking, sitting, and interacting with their environment from a occupational therapist point of view.

Study Design:

Participants will be divided into three distinct groups:

1. Group 1: Deaf children with confirmed vestibular impairment.
2. Group 2: Deaf children without vestibular impairment.
3. Group 3 (Control Group): Hearing children without vestibular deficits. A total of 105 children (35 per group) will be enrolled over a three-year period during their consultations at the ENT departement.

Methods and Data Collection:

• Quantitative Evaluation:

Children's daily life activities will be assessed using the OT Hope 0-5 years questionnaire, which is completed by parents with assistance from an occupational therapist. This tool measures children's competences across key domains, including personal care, play, and social interactions. Responses are categorized into four levels:

* ""Yes, we can do this.""
* ""Yes, we can do this with help.""
* ""We can't do this very well.""
* ""No, we can't do this."" Scores will be assigned to each response, and the overall scores will be compared between the three groups to identify differences in competences and daily activity performance.

  * Qualitative Evaluation:

It will be proposed to some parents to participate in qualitative interviews designed to explore their experiences, challenges, and strategies related to their child's daily routines and motor development. These interviews will provide insights on the impact of vestibular impairments on family life and the child's autonomy.

Hypotheses:

The study is based on the following hypotheses:

1. Deaf children with vestibular impairments will have lower scores in daily life activities, especially in motor-related tasks such as walking, compared to the other two groups.
2. Deaf children without vestibular impairments may show slight differences compared to hearing children due to their hearing loss but will perform better than children with both hearing and vestibular impairments.
3. The qualitative interviews will reveal specific challenges faced by families of children with vestibular dysfunction and highlight adaptive strategies.

Outcomes:

* Primary Outcome: Comparison of daily life activity scores between the three groups using the OT Hope 0-5 years tool.
* Secondary Outcomes: Analysis of qualitative interview data to explore themes related to motor challenges, family adaptation, and participation in daily routines.

Study Duration:

* Inclusion period: 3 years.
* Patient participation: Approximately 1 hour (including questionnaire completion and, for some, qualitative interviews).

Ethical and Regulatory Considerations:

The study complies with ethical standards for human research and data confidentiality regulations. Parents' non-opposition will be documented, and all collected data will be anonymized and securely stored.

By exploring both quantitative and qualitative dimensions, this study aims to provide a comprehensive understanding of how vestibular impairments affect the functional development and autonomy of young children, with the ultimate goal of guiding early interventions and improving clinical practices.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Deaf children with confirmed vestibular impairment. Group 2: Deaf children without vestibular impairment. Group 3: Hearing children without vestibular impairment (control group).

Exclusion Criteria:

Presence of neuromotor or orthopedic disorders. Presence of pervasive developmental disorders that could interfere with daily activity assessments."

Ages: 1 Day to 2 Years | Sex: All
Age Groups: Child
Study Population: Children coming in consultations in the ENT department
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-03-27 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
OT Hope 0 - 5 ans Therapeutic tool for self determination of pediatric goals in occupational therapy | 15 minutes
  Assessment of daily life activities in children aged 0-2 years using the OT Hope 0-5 tool. Parents rate their child's performance in personal care, play, and social interactions. Scores associated will be compared across three groups to evaluate the impact of vestibular impairments.

SECONDARY OUTCOMES:
Qualitative interviews with parents | 45 minutes
  Exploration of parents' perspectives through qualitative interviews to understand how vestibular impairments affect their child's daily life activities, challenges encountered, and strategies used to support participation.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MAUDOUX, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided